CLINICAL TRIAL: NCT04694599
Title: The Effect of Continuous Pulse Oximetry Monitoring and Early Intervention Using Wearable Device on the Incidence of Postoperative Hypoxemia a Randomized Controlled Trial
Brief Title: The Effect of Continuous Pulse Oximetry Monitoring and Early Intervention Using Wearable Device on the Incidence of Postoperative Hypoxemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RadiusPPG
Record Dates: First submitted 2021-01-03; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Respiratory Complication

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Early intervention (Experimental): The experimental group will receive oxygen supplementation when oxygen saturation decreases according to the monitoring of wearable devices.
  Interventions: Device: Low flow oxygen
- Typical (Active Comparator): The control group will receive oxygen supplementation when oxygen saturation decreases according to typical periodical monitoring.
  Interventions: Device: Low flow oxygen

INTERVENTIONS:
Device: Low flow oxygen — Low flow oxygen delivered via nasal prong or facial mask. The flow rate is adjusted according to oxygen saturation of the patient.

SUMMARY:
Vital signs of postoperative patient are monitored intensively in post-anesthesia care unit or intensive care unit, but the frequency of surveillance decreases in typical surgical wards. The continuous pulse oximetry in surgical wards is known to be useful in detection and prevention of hypoxemia, reducing complications caused by postoperative respiratory depression. However, continuous monitoring is not conducted, due to shortage of equipment and personnel. Recently, wearable device for measuring pulse oxygen saturation, which is inexpensive, applicable to patients with mobility, and can be monitored continuously through wireless connection, has been supplied. In this study, the investigators evaluate the effect of continuous monitoring of oxygen saturation with wireless device(MASIMO Radius-7) on postoperative patients who are transferred to general wards, and evaluate the effect of early intervention in reducing the event of hypoxemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing noncardiac surgery under general anesthesia
* American Society of Anesthesiologists (ASA) physical status class I-III

Exclusion Criteria:

* Patients refusing to participate in the study
* Patients under emergency surgery
* Patients who wearable device is not applicable
* Patients scheduled to be transferred to intensive care unit
* Patients scheduled to receive oxygen supplementation in surgical ward
* Patients scheduled to undergo continuous pulse oximetry monitoring

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
The prevalence of prolonged hypoxemic episodes | 24 hours after transfer to surgical ward
  the prevalence of hypoxia lasting more than 1 hour, according to a threshold of SpO2<90%

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun Z, Sessler DI, Dalton JE, Devereaux PJ, Shahinyan A, Naylor AJ, Hutcherson MT, Finnegan PS, Tandon V, Darvish-Kazem S, Chugh S, Alzayer H, Kurz A. Postoperative Hypoxemia Is Common and Persistent: A Prospective Blinded Observational Study. Anesth Analg. 2015 Sep;121(3):709-715. doi: 10.1213/ANE.0000000000000836. PMID 26287299
- [Background] Ishikawa M, Sakamoto A. Postoperative desaturation and bradypnea after general anesthesia in non-ICU patients: a retrospective evaluation. J Clin Monit Comput. 2020 Feb;34(1):81-87. doi: 10.1007/s10877-019-00293-0. Epub 2019 Mar 2. PMID 30827008
- [Background] Ramachandran SK, Thompson A, Pandit JJ, Devine S, Shanks AM. Retrospective observational evaluation of postoperative oxygen saturation levels and associated postoperative respiratory complications and hospital resource utilization. PLoS One. 2017 May 17;12(5):e0175408. doi: 10.1371/journal.pone.0175408. eCollection 2017. PMID 28520718
- [Background] Weenk M, Bredie SJ, Koeneman M, Hesselink G, van Goor H, van de Belt TH. Continuous Monitoring of Vital Signs in the General Ward Using Wearable Devices: Randomized Controlled Trial. J Med Internet Res. 2020 Jun 10;22(6):e15471. doi: 10.2196/15471. PMID 32519972
- [Background] Breteler MJM, KleinJan EJ, Dohmen DAJ, Leenen LPH, van Hillegersberg R, Ruurda JP, van Loon K, Blokhuis TJ, Kalkman CJ. Vital Signs Monitoring with Wearable Sensors in High-risk Surgical Patients: A Clinical Validation Study. Anesthesiology. 2020 Mar;132(3):424-439. doi: 10.1097/ALN.0000000000003029. PMID 31743149